CLINICAL TRIAL: NCT02121535
Title: Bioequivalence of Telmisartan 80 mg/Amlodipine 5 mg/Hydrochlorothiazide 12.5 mg Fixed-dose Combination Tablet Compared to Concomitant Administration of Telmisartan 80 mg/Amlodipine 5 mg Fixed-dose Combination Tablet and Hydrochlorothiazide 12.5 mg Tablet in Healthy Male Subjects : an Open-label, Randomised, Single-dose, Two-sequence, Four-period Replicated Crossover Study
Brief Title: Bioequivalence Study of Telmisartan Between T80/A5/H12.5 mg FDC Tablet and T80/A5 mg Tab and H12.5 mg Tab Concomitant Use
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1348.3
Record Dates: First submitted 2014-04-22; First posted 2014-04-23 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Healthy

ARMS (2):
- T80/A5/H12.5 mg FDC (Experimental): A Telmisartan 80 mg/Amlodipine 5 mg/Hydrochlorothiazide 12.5 mg fixed dose combination (FDC) tablet
  Interventions: Drug: T80/A5 mg FDC tablet; Drug: H12.5 mg tablet; Drug: T80/A5/H12.5 mg FDC tablet
- T80/A5 mg FDC+H12.5 mg mono (Active Comparator): A Telmisartan 80 mg/ Amlodipine 5 mg fixed dose combination (FDC) tablet and a Hydrochlorothiazide 12.5 mg tablet
  Interventions: Drug: T80/A5 mg FDC tablet; Drug: T80/A5/H12.5 ng FDC tablet; Drug: H12.5 mf tablet

INTERVENTIONS:
Drug: T80/A5 mg FDC tablet
  Arms: T80/A5/H12.5 mg FDC
Drug: T80/A5 mg FDC tablet — A Telmisartan 80 mg/ Amlodipine 5 mg FDC tablet
  Arms: T80/A5 mg FDC+H12.5 mg mono
Drug: H12.5 mg tablet
  Arms: T80/A5/H12.5 mg FDC
Drug: T80/A5/H12.5 ng FDC tablet — A Telmisartan 80 mg/Amlodipine 5 mg/HCTZ 12.5 mg FDC tablet
  Arms: T80/A5 mg FDC+H12.5 mg mono
Drug: H12.5 mf tablet — A HCTZ 12.5 mg tablet
  Arms: T80/A5 mg FDC+H12.5 mg mono
Drug: T80/A5/H12.5 mg FDC tablet
  Arms: T80/A5/H12.5 mg FDC

SUMMARY:
The study will be performed as an open-label, randomised, single-dose, two-sequence, four-period replicated crossover design. A total of 72 Japanese healthy male subjects will be randomised to 2 groups. The subjects are administrated either T80/A5/H12.5 mg FDC tablet once or T80/A5 mg FDC tablet and hydrochlorothiazide (HCTZ) 12.5 mg tablet once in each period. The length of admission will be 7 days in each period.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects age =20 and =35 years; body weight: =50 kg and =80 kg; body mass index: =18.0 and =25.0 kg/m2
* Without any clinically significant findings and complications on the basis of a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR), body temperature), 12-lead electrocardiograms (ECGs), clinical laboratory tests
* Signed and dated written informed consent prior to admission to the trial in accordance with the Good Clinical Practice (GCP) and the local legislation.

Exclusion criteria:

- Any finding of the medical examination (including BP, PR and ECGs) deviating from normal and of clinical relevance.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Boehringer Ingelheim Investigational Site, Kanagawa, Yokohama, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was performed as an open-label, randomised, single-dose, two-sequence, four period replicated crossover design. A total of 72 healthy male subjects were randomised to 2 groups (Treatment sequences 1 or 2).
Groups:
- Sequence TRRT: Oral administration of study drugs in the following order: T (period 1) - R(period 2) - R (period 3) - T (period 4).
  T: telmisartan 80mg+amlodipine 5mg+ hydrochlorothiazide (HCTZ) 12.5mg fix dose tab, once daily; R: telmisartan 80mg+amlodipine 5mg fixed dose combination (FDC) + HCTZ 12.5mg tablet , once daily.
  The washout period between drug administrations had to be at least 14 days from the study drug administration of the previous period.
- Sequence RTTR: Oral administration of study drugs in the following order: R (period 1) - T (period 2) - T (period 3) - R (period 4).
  T: telmisartan 80mg+amlodipine 5mg+HCTZ 12.5mg fix dose tab, once daily; R: telmisartan 80mg+amlodipine 5mg FDC + HCTZ 12.5mg tablet , once daily. The washout period between drug administrations had to be at least 14 days from the study drug administration of the previous period.
Period: Period 1 (8 Trial Days)
Arm/Group | Sequence TRRT | Sequence RTTR
Started | 36 | 36
Completed | 36 | 35 (1 subject withdrew his consent during the washout period between Period 1 and 2.)
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Period 2 (8 Trial Days)
Arm/Group | Sequence TRRT | Sequence RTTR
Started | 36 | 35
Completed | 36 | 35
Not Completed | 0 | 0
Period: Period 3 (8 Trial Days)
Arm/Group | Sequence TRRT | Sequence RTTR
Started | 36 | 35
Completed | 35 (1 subject withdrew consent during the washout period between Period 3 and 4.) | 35
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 4 (8 Trial Days)
Arm/Group | Sequence TRRT | Sequence RTTR
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): TS included all subjects who were dispensed with the study drugs and were documented to have taken at least 1 dose of the study drugs. Safety analyses were conducted on the TS.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sequence TRRT | Sequence RTTR | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.3 (4.7) | 27.2 (5.0) | 26.7 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 36 | 36 | 72

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of the Telmisartan in Plasma Over the Time Interval From 0 to the Time of the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the telmisartan in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz)
Time Frame: 3hours(h) before drug administration and 15minutes (m), 30m, 45m, 1h, 1h30m, 2h, 2h30m, 3h, 4h, 6h, 8h, 12h, 24h, 32h, 48h, 72h after drug administration
Population: Pharmacokinetic set (PKS):
  included all subjects in the TS who had evaluable pharmacokinetic (PK) variables for both test drug and reference drugs. Subjects who had an important protocol violation (PV) for relevant PK evaluation were excluded from the PKS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Test Treatment: Oral administration of telmisartan 80mg+amlodipine 5mg+HCTZ 12.5mg fixed dose combination (FDC), once daily;
- Reference Treatment: Oral administration of telmisartan 80mg+amlodipine 5mg FDC + HCTZ 12.5mg tablet , once daily.
Arm/Group | Test Treatment | Reference Treatment
Number analyzed (Participants) | 71 | 71
ng*h/mL | 2850 (52.0) | 2790 (54.9)
Statistical Analysis 1: Comparison: Test Treatment vs Reference Treatment; The statistical model used for the analysis of AUC0-tz was a mixed effect model on the logarithmic scale; Test type: Non-Inferiority or Equivalence — To determine whether the 2-sided 90% confidence interval (CI) for the intra-subject ratio of the AUC0-tz were contained in the acceptance range of 80% to 125% for bioequivalence; Adjusted Mean Ratio = 101.97, 90% CI 2-sided [98.94 to 105.08] — Adjusted Mean Ratio (Test/Reference)

2. Primary Outcome: Cmax for Telmisartan
Description: Cmax (maximum measured concentration of the analyte in plasma)
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Test Treatment | Reference Treatment
Number analyzed (Participants) | 71 | 71
ng/mL | 718 (56.4) | 694 (55.2)
Statistical Analysis 1: Comparison: Test Treatment vs Reference Treatment; The statistical model used for the analysis of Cmax was a mixed effect model on the logarithmic scale; Test type: Non-Inferiority or Equivalence — To determine whether the 2-sided 90% CI for the intra-subject ratio of the Cmax were contained in the acceptance range of 80% to 125% for bioequivalence; Adjusted Mean Ratio = 103.77, 90% CI 2-sided [97.03 to 110.99] — Adjusted Mean Ratio (Test/Reference)

3. Secondary Outcome: AUC0-∞ for Telmisartan
Description: AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Test Treatment | Reference Treatment
Number analyzed (Participants) | 71 | 71
ng*h/mL | 3090 (54.5) | 3120 (58.8)
Statistical Analysis 1: Comparison: Test Treatment vs Reference Treatment; The statistical model used for the analysis of AUC0--∞ was a mixed effect model on the logarithmic scale; Test type: Non-Inferiority or Equivalence — To determine whether the 2-sided 90% CI for the intra-subject ratio of the AUC0-∞ were contained in the acceptance range of 80% to 125% for bioequivalence; Adjusted Mean Ratio = 100.24, 90% CI 2-sided [96.80 to 103.80] — Adjusted Mean Ratio (Test/Reference)

4. Secondary Outcome: AUC0-∞ for Amlodipine
Description: as for outcome 3
Time Frame: 3hours(h) before drug administration and 1h, 2h, 3h, 4h, 6h, 8h, 12h, 24h, 32h, 48h, 72h, 96h, 120h, 144h after drug administration
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Test Treatment | Reference Treatment
Number analyzed (Participants) | 71 | 71
ng*h/mL | 184 (25.2) | 185 (26.0)
Statistical Analysis 1: Comparison: Test Treatment vs Reference Treatment; The statistical model used for the analysis of AUC0--∞ was a mixed effect model on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Adjusted Mean Ratio = 99.42, 90% CI 2-sided [97.94 to 100.93] — Adjusted Mean Ratio (Test/Reference)

5. Primary Outcome: AUC0-tz for Amlodipine
Description: AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point)
Time Frame: as for outcome 4
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Test Treatment | Reference Treatment
Number analyzed (Participants) | 71 | 71
ng*h/mL | 171 (24.3) | 172 (25.0)
Statistical Analysis 1: Comparison: Test Treatment vs Reference Treatment; The statistical model used for the analysis of AUC0-tz was a mixed effect model on the logarithmic scale; Test type: Non-Inferiority or Equivalence — To determine whether the 2-sided 90% CI for the intra-subject ratio of the AUC0-tz were contained in the acceptance range of 80% to 125% for bioequivalence; Adjusted Mean Ratio = 99.50, 90% CI 2-sided [98.08 to 100.94] — Adjusted Mean Ratio (Test/Reference)

6. Primary Outcome: Cmax for Amlodipine
Description: Cmax (maximum measured concentration of the analyte in plasma)
Time Frame: as for outcome 4
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Test Treatment | Reference Treatment
Number analyzed (Participants) | 71 | 71
ng/mL | 3.69 (22.0) | 3.68 (20.7)
Statistical Analysis 1: Comparison: Test Treatment vs Reference Treatment; The statistical model used for the analysis of Cmax was a mixed effect model on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Adjusted Mean Ratio = 100.07, 90% CI 2-sided [98.45 to 101.72] — Adjusted Mean Ratio (Test/Reference)

7. Primary Outcome: Cmax for Hydrochlorothiazide
Description: Cmax (maximum measured concentration of the analyte in plasma)
Time Frame: 3hours(h) before drug administration and 15minutes (m), 30m, 45m, 1h, 1h30m, 2h, 2h30m, 3h, 4h, 6h, 8h, 12h, 24h, 32h, 48h after drug administration
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Test Treatment | Reference Treatment
Number analyzed (Participants) | 71 | 71
ng/mL | 104 (23.0) | 94.7 (23.4)
Statistical Analysis 1: Comparison: Test Treatment vs Reference Treatment; The statistical model used for the analysis of Cmax was a mixed effect model on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Adjusted Mean Ratio = 110.16, 90% CI 2-sided [106.87 to 113.54] — Adjusted Mean Ratio (Test/Reference)

8. Primary Outcome: AUC0-tz for Hydrochlorothiazide
Description: as for outcome 5
Time Frame: as for outcome 7
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Test Treatment | Reference Treatment
Number analyzed (Participants) | 71 | 71
ng*h/mL | 638 (19.3) | 611 (19.6)
Statistical Analysis 1: Comparison: Test Treatment vs Reference Treatment; The statistical model used for the analysis of AUC0-tz was a mixed effect model on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 5, analysis 1]; Adjusted Mean Ratio = 104.30, 90% CI 2-sided [102.53 to 106.10] — Adjusted Mean Ratio (Test/Reference)

9. Secondary Outcome: AUC0-∞ for Hydrochlorothiazide
Description: as for outcome 3
Time Frame: as for outcome 7
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Test Treatment | Reference Treatment
Number analyzed (Participants) | 71 | 71
ng*h/mL | 661 (18.7) | 634 (18.9)
Statistical Analysis 1: Comparison: Test Treatment vs Reference Treatment; The statistical model used for the analysis of AUC0--∞ was a mixed effect model on the logarithmic scale; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Adjusted Mean Ratio = 104.37, 90% CI 2-sided [102.68 to 106.10] — Adjusted Mean Ratio (Test/Reference)

ADVERSE EVENTS:
Time Frame: Adverse Events occurring after the first study drug administration till the end of treatment (EOT) (EOT: 144 hours after drug administration)
Groups:
- Total (All Patients): Total of all the participants analyzed
Arm/Group | Test Treatment | Reference Treatment | Total (All Patients)
Serious Adverse Events (participants affected / at risk) | 0/71 | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 0/71 | 0/72 | 0/72

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights